CLINICAL TRIAL: NCT00862914
Title: Immunohistochemical Expression Patterns of microRNA Processing Enzyme Dicer in Cutaneous Malignant Melanoma, Benign and Dysplastic Melanocytic Naevi
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Dr., Ruhr University of Bochum
Other Study IDs: 006
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Naevi; Malignant Melanoma
Keywords: Skin; MicroRNA; miRNA; Dicer; Malignant Melanoma
MeSH Terms: conditions — Nevus; Melanoma; Rhabdomyosarcoma, Embryonal, 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paraffin embedded melanocytic skin lesion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: benign melanocytic naevi
- 2: dysplastic melanocytic naevi
- 3: cutaneous malignant melanoma

SUMMARY:
MicroRNAs (miRNAs) are very small endogenous RNA molecules about 22-25 nucleotides in length, capable of post-transcriptional gene regulation. miRNAs bind to their target messenger RNAs (mRNAs), leading to cleavage or suppression of target mRNA translation based on the degree of complementarity. miRNAs have recently been shown to play pivotal roles in diverse developmental and cellular processes and linked to a variety of skin diseases and cancers. In the present study the researchers investigate the immunohistochemical distribution of Dicer in benign and dysplastic melanocytic naevi as well as in cutaneous malignant melanoma compared to intraindividual healthy control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign melanocytic naevi, dysplastic melanocytic naevi and cutaneous malignant melanoma.

Exclusion Criteria:

* Patients under 18 years of age
* Patients with other forms of cancer in previous medical history
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dermatologic primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Peter Altmeyer, Principal Investigator — Department of Dermatology and Allergology, Ruhr-University Bochum; PD Dr. Falk G. Bechara, Study Director — Department of Dermatology and Allergology, Ruhr-University Bochum
Locations (1):
- Department of Dermatology and Allergology, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Gambichler T, Sand D, Altmeyer P, Stuecker M, Bechara FG. Immunohistochemical expression patterns of the microRNA-processing enzyme Dicer in cutaneous malignant melanomas, benign melanocytic nevi and dysplastic melanocytic nevi. Eur J Dermatol. 2011 Jan-Feb;21(1):18-21. doi: 10.1684/ejd.2011.1210. PMID 21262599